CLINICAL TRIAL: NCT06665750
Title: Effect of Neuromuscular Training on Upper Extremity Performance in Recreational Tennis Players
Brief Title: Neuromuscular Training in Recreational Tennis Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Meltem Koc, Assist Prof, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 230155/24
Record Dates: First submitted 2024-10-20; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Sport Injuries
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: Exercise
- Control group (No Intervention): The control group will perform only routine warm-up exercises.

INTERVENTIONS:
Behavioral: Exercise — A progressive upper extremity neuromuscular exercise program was performed face to face with the researcher physiotherapist for the study group. The exercise program was applied for approximately 20 minutes, 2 days a week for 6 weeks, on the same days of the week, before the participants' tennis training. The exercise content and number of repetitions in the training program changed every 2 weeks with increasing difficulty.
  Arms: Intervention group

SUMMARY:
The aim of this study is to investigate the effect of upper extremity neuromuscular exercise training on throwing performance, upper extremity strength, and endurance in recreational tennis players. In this context, 24 recreational tennis players will be included in the study. Participants will be divided into two equal groups using a simple randomization method. The study group (n=12) will receive progressive upper extremity neuromuscular exercise training twice a week for six weeks before each tennis training session, while the control group will perform only routine warm-up exercises. Both groups will be evaluated twice, once at the beginning of the study and again at the end of the six-week intervention. Throwing performance will be assessed using the Functional Throwing Performance Index (FTPI) and the International Tennis Number Test (ITN). Upper extremity endurance will be evaluated through the Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST) and Scapula Muscle Endurance Test (SME), while upper extremity strength will be measured using the Health Ball Throw Test (HBT) and the Y Balance Upper Extremity Test (YBUET). Statistical analysis will be conducted using SPSS 24.0 software.

ELIGIBILITY:
Inclusion Criteria:

1. Being between the ages of 18-50
2. Being a recreational tennis player
3. Playing tennis regularly for at least 1 year
4. Playing tennis regularly at least twice a week for the last 6 months

Exclusion Criteria:

1. Playing another sport along with tennis
2. Being a professional tennis player
3. Having a history of any injury and/or surgery affecting the upper extremity

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Functional Throwing Performance Index (FTPI) | baseline and after six weeks

SECONDARY OUTCOMES:
International Tennis Number Test (ITN) | baseline and after six weeks
Closed Kinetic Chain Upper Extremity Stability Test | Baseline and after six weeks
Scapula Muscle Endurance Test | Baseline and after six weeks
Health Ball Throw Test | Baseline and after six weeks
Y Balance Upper Extremity Test | Baseline and after six weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Mugla Sitki Kocman University, Menteşe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No